CLINICAL TRIAL: NCT04197154
Title: Pain-related Fear as a Facilitator of Nocebo Hyperalgesia: An Experimental Study
Brief Title: Pain-related Fear as a Facilitator of Nocebo Hyperalgesia
Acronym: LFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Universiteit Leiden (Other); KU Leuven (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, AWMEvers, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CEP19-0614/347
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Hyperalgesia; Chronic Pain Syndrome; Chronic Pain, Psychogenic; Fear of Pain
Keywords: Nocebo; Pain; Fear; Conditioning; Negative suggestions; Extinction
MeSH Terms: conditions — Hyperalgesia; Chronic Pain; Pain | interventions — Extinction, Biological

STUDY DESIGN:
Who Masked: Participant
Masking Description: A double-blind randomization list (stratified for gender) was created by an independent researcher. Complete blinding of the researchers during the experiment is not possible due to the nature of the conditioning paradigms. However, in this study blinding is optimized: the researchers are informed of the (conditioning) group to which participants are allocated after their final inclusion to the study and after the start of the experiment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Control nocebo group (Experimental): Conditioning and extinction of a nocebo response using moderate pain stimuli, nocebo negative suggestions, and no threat suggestions.
  Interventions: Behavioral: Threat manipulation (control, no threat); Behavioral: Conditioning of moderate pain; Behavioral: Extinction
- 2. High-pain nocebo group (Experimental): Conditioning and extinction of a nocebo response using higher pain stimuli, nocebo negative suggestions, and no threat suggestions.
  Interventions: Behavioral: Threat manipulation (control, no threat); Behavioral: Conditioning of high pain; Behavioral: Extinction
- 3. High-threat nocebo (Experimental): Conditioning and extinction of a nocebo response using moderate pain stimuli, nocebo negative suggestions, and threat suggestions (i.e., fear-inducing suggestions).
  Interventions: Behavioral: Threat manipulation; Behavioral: Conditioning of moderate pain; Behavioral: Extinction

INTERVENTIONS:
Behavioral: Threat manipulation (control, no threat) — Before the start of conditioning, a mock skin-sensitivity test informs participants that their skin reacts to heat normally and it is safe for them to participate. A skin-sensitivity reading shows participants a scale that is in the green (no danger) zone.
  Arms: 1. Control nocebo group; 2. High-pain nocebo group
Behavioral: Threat manipulation — Before the start of conditioning, a mock skin-sensitivity test informs participants that their skin is very sensitive and their nerve fibers are very responsive and they may have adverse reactions to the heat-pain application. A skin-sensitivity reading shows participants a scale that is in the red (higher danger) zone.
  Arms: 3. High-threat nocebo
Behavioral: Conditioning of moderate pain — During nocebo trials of the acquisition phase, conditioned stimuli (i.e., on-screen visual cues "ON" signaling the activation of sham electrical stimulation) are paired to unconditioned moderate-pain stimuli, to induce a negative association between the activation of electrical stimuli and an increase in pain. During control trials of the acquisition phase, the deactivation of the sham electrical stimulation (i.e., on-screen message "OFF") is paired to 'baseline' pain of lower intensity.
  Other Names: Nocebo Induction
  Arms: 1. Control nocebo group; 3. High-threat nocebo
Behavioral: Conditioning of high pain — During nocebo trials of the acquisition phase, conditioned stimuli (i.e., on-screen visual cues "ON" signaling the activation of sham electrical stimulation) are paired to unconditioned high-pain stimuli, to induce a negative association between the activation of electrical stimuli and an increase in pain. During control trials of the acquisition phase, the deactivation of the sham electrical stimulation (i.e., on-screen message "OFF") is paired to pain of lower intensity.
  Other Names: Nocebo Induction
  Arms: 2. High-pain nocebo group
Behavioral: Extinction — During extinction, the previously conditioned nocebo effects on pain are attenuated by pairing the nocebo and control visual cues (i.e., on-screen messages "ON" and "OFF") to pain stimuli of only lower intensity.
  Other Names: Nocebo Attenuation

SUMMARY:
Nocebo hyperalgesia is characterized by adverse pain outcomes, induced by patients' expectations. In the lab, nocebo effects are commonly studied via classical conditioning, a method that employs pairings of neutral cues/treatments with different pain intensities to install differential pain-related expectations. In such conditioning experiments, participants are typically taught that a (sham) treatment exaggerates their pain, by surreptitiously administering high intensity (e.g. pain) stimuli in combination with this treatment. Verbal suggestions are also often used to inform participants of the supposed adverse effects of such treatments. In nocebo studies, higher pain levels and suggestions that are of more threatening nature may induce fear, thereby adding a crucial element to the experimental manipulation. Since nocebo effects are hypothesized to arise in clinical settings due to a combination of several psychological and cognitive mechanisms, it is important to study the role that factors such as higher pain levels, conditioned pain-related fear, or more threatening verbal suggestions may play in the formation of nocebo hyperalgesia. To date, no studies have focused on the fear-inducing effect that different pain intensities or verbal threat suggestions may have and how this fear, in turn, may strengthen the acquisition of nocebo effects. This study aims to investigate whether higher pain intensity or higher pain-related fear induced via threatening suggestions facilitate the acquisition and hinder subsequent extinction of nocebo hyperalgesia. This study will be conducted at Leiden University.

DETAILED DESCRIPTION:
The investigators expect that higher pain intensity and/or higher pain-related fear induced via threatening suggestions will lead to stronger acquisition of nocebo hyperalgesia and/or more durable nocebo hyperalgesia after extinction.

Main outcome variables:

* The magnitude of induced nocebo hyperalgesia is defined as the difference in pain ratings for the first nocebo trial compared to the first control trial of the extinction phase.
* The reduction of nocebo hyperalgesia is defined as the change in reported pain between the first and last nocebo trial of the extinction phase.
* Fear levels (for mediation analyses) are measured via eye-blink startle modulation and self-reported fear during nocebo trials (relative to control trials).

For EMG analyses this study follows typical pre-processing of EMG recordings, similar to previous studies. The EMG signal will be digitized at 1,000 Hz from 200 ms before the startle probe until 1,500 ms after probe onset. The startle probe is a 100 dBA burst of white noise with instantaneous rise time presented binaurally for 100 ms through earphones. Each 2-4 consecutive startle probe responses of the same cue (nocebo vs control) will be averaged for further analyses. Participants who exhibited a startle response in less than 20% of trials in the first half of induction will be labeled as non-responders. Trials during which, for example, baseline is higher than startle response peak due to an occasional blink before the probe presentation, will be labelled as non-response or reject trials.

1. Main planned analyses:

   To examine whether higher pain stimulation (high-pain nocebo group) leads to stronger nocebo hyperalgesia, as compared to lower pain stimulation (control nocebo group), a 2x2 mixed model analysis of variance (ANOVA) will be performed with group (high-pain nocebo group, control nocebo group) as the between-subjects factor and trial type as within-subjects factor with two levels (first nocebo extinction trial, first control extinction trial).
2. Secondary analyses:

2a. To examine whether an impact of higher pain stimulation on the magnitude of nocebo hyperalgesia was mediated by pain-related fear levels, a mediation analysis will be conducted for the high pain nocebo and control nocebo groups, to assess if fear mediates the relationship between pain levels and the magnitude of nocebo hyperalgesia (calculated difference scores between the first nocebo extinction trial and the first control extinction trial).

2b. To examine whether higher pain-related fear induced via a threat suggestion (high-threat nocebo) led to stronger nocebo hyperalgesia, as compared to no threat suggestion (control nocebo group), a 2x2 mixed model ANOVA will be performed with group (high-threat nocebo, control nocebo group) as the between-subjects factor and trial type as within-subjects factor with two levels (first nocebo extinction trial, first control extinction trial).

2c. To examine whether higher pain stimulation (high-pain nocebo group) led to more durable nocebo effect, as compared to lower pain stimulation (control nocebo group), a 2x2 mixed model ANOVA will be performed with group (high-pain nocebo group, control nocebo group) as the between-subjects factor and trial as within-subjects factor with two levels (first nocebo extinction trial, last nocebo extinction trial).

2d. To examine whether an impact of higher pain stimulation on the durability of nocebo hyperalgesia was mediated by pain-related fear levels, a mediation analysis will be conducted to assess if fear mediates the relationship between pain levels and the magnitude of nocebo hyperalgesia after extinction (calculated difference scores between the first nocebo extinction trial and the last nocebo extinction trial).

2e. To examine whether higher pain-related fear induced via a threat suggestion led to more durable nocebo hyperalgesia, as compared to no threat suggestion, a 2x2 mixed model ANOVA will be performed with group (high-threat nocebo, control nocebo group) as the between-subjects factor and trial as within-subjects factor with two levels (first nocebo extinction trial, last nocebo extinction trial).

ELIGIBILITY:
Inclusion Criteria:

* Aged 17 - 35 years
* Good understanding of the English language
* Normal or corrected to normal vision

Exclusion Criteria:

* Ever having experienced serious medical or psychiatric conditions (e.g., heart or lung disease, panic attacks, drug addiction, clinical depression),
* Ever having experienced chronic pain complaints (pain for more than 6 months),
* Experiencing acute physical pain (e.g., headache; above 3 on a 10-point NRS scale), or having used pain medication on the day of testing,
* Pregnancy or breastfeeding,
* Having recent injuries to the wrists or arms on the day of testing,
* Previous participation in this or similar studies (e.g., using conditioning or thermal pain).
* Having consumed psychotropic medication, recreational drugs, analgesic medication, or more than 3 units of alcohol, in the 24 hours prior to the study appointment.
* After inclusion, participants who do not reach a sensation of high pain (at least 6 on the NRS) with the highest administered temperature or participants who appear unable to distinguish between moderate and high pain stimuli (reporting at least a mean difference of 1.5 NRS points between nocebo and control trials during induction) will also be excluded.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants whose lived gender is male, will be included as male and participants whose lived gender is female, will be included as female.
Enrollment: 72 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Magnitude of nocebo hyperalgesia | On the testing day, in the first trials of the extinction phase
  The magnitude of induced nocebo hyperalgesia is defined as the difference in pain ratings for the first nocebo trial compared to the first control trial of the extinction phase.

SECONDARY OUTCOMES:
Reduction of nocebo hyperalgesia | On the testing day, in the extinction phase
  The reduction of nocebo hyperalgesia is defined as the change in reported pain between the first and last nocebo trial of the extinction phase.

OTHER OUTCOMES:
Fear levels | On the testing day, in both experimental phases
  Fear levels (for mediation analyses) are measured via eye-blink startle modulation
Fear self report levels | On the testing day, in both experimental phases
  Fear levels (for mediation analyses) are also measured via self-reported fear during nocebo trials (relative to control trials).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea WM Evers, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All data are collected pseudonymised; consent forms are the only sources containing personal data and will not be shared, but are monitored by the department's Data Monitor.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available immediately after publication of the study and will be retained for 15 years.
Access Criteria: Data can be shared with scientists in relevant fields for the purpose of future studies such as replication or meta-analysis (or with designated persons for monitoring purposes).